CLINICAL TRIAL: NCT03310567
Title: A Phase 2 Study of Pembrolizumab in Combination With Epacadostat in Women With Recurrent/Metastatic Endometrial Carcinoma
Brief Title: A Study of Pembrolizumab in Combination With Epacadostat in Women With Recurrent/Metastatic Endometrial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsors pulled out of the study
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN-104
Record Dates: First submitted 2017-10-06; First posted 2017-10-16 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Recurrent/ Metastatic Endometrial Carcinoma
MeSH Terms: interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Women with recurrent/ metastatic endometrial carcinoma would be treated with Epacadostat and pembroluzimab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epacadostat + pembrolizumab (Experimental)
  Interventions: Drug: Epacadostat + pembrolizumab

INTERVENTIONS:
Drug: Epacadostat + pembrolizumab — Each patient would be administered epacadostat orally twice a day and pembroluzimab by infusion once in a cycle of 21 days

SUMMARY:
Expression of IDO and PD-1/L1 has been found to be increased in endometrial cancer. Expression of these markers on the tumor cells leads to immunosuppression in the micro-environment of tumors that prevents immune system from attacking and killing tumor cells. The purpose of this trial is to target these antigens by concomitant administration of drugs epacadostat and pembrolizumab, thereby removing twin mechanisms of immune-suppression that may lead to better control of tumor growth.

DETAILED DESCRIPTION:
Primary Objective

* Evaluate the response rate (RR) and 6 month progression-free survival (PFS-6) of patients with recurrent or metastatic endometrial carcinoma when treated with epacadostat in combination with pembrolizumab as measured by modified RECIST v1.1
* In a subset analysis, evaluate the response rate (RR) and 6 month progression-free survival (PFS-6) of patients with microsatellite instability (MSI) and recurrent or metastatic endometrial carcinoma when treated with epacadostat in combination with pembrolizumab.

Secondary Objectives

* Evaluate the safety and tolerability of epacadostat in combination with pembrolizumab.
* Evaluate the overall survival (OS) of patients with recurrent or metastatic endometrial carcinoma when treated with epacadostat in combination with pembrolizumab as measured by modified RECIST v1.1.
* In a subset analysis, evaluate the overall survival (OS) of patients with microsatellite instability (MSI) and recurrent or metastatic endometrial carcinoma when treated with epacadostat in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign an informed consent form (ICF).
* Women aged 18 years or older.
* Subjects must have histologically confirmed diagnosis of endometrial cancer, which is recurrent, persistent or metastatic.
* Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, mixed epithelial carcinoma and carcinosarcoma (MMMT)
* Presence of measurable disease per RECIST v1.1
* Patients must have archived tissue specimen not more than 10 years old.
* Subjects must have an ECOG performance status of 0 or 1.
* Patients must have recovered (ie, grade ≤1 toxicity or patient's baseline status, except alopecia) from all previous treatment-related toxicities.
* Prior therapy must include platinum and taxane combination therapy.
* Patients must have recurrence or progression of disease after one line of therapy in the metastatic/recurrent setting
* Life expectancy >12 weeks
* Patients must have normal organ and marrow functions as defined below. All screening laboratory tests should be performed within 7 days of treatment initiation System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L (transfusion is acceptable to meet this criteria) Renal Serum creatinine OR Measured or calculated a creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

  * 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ ULN OR If total bilirubin exceeds the ULN, conjugated bilirubin must be checked, and subjects should be excluded if the value is above the ULN.

AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

* Female participants of childbearing potential must have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication. They should also be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Refer to section 4.4 for more details. All female subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through 120 days after the last dose of study treatment. Permitted methods that are at least 99% effective in preventing pregnancy. See Appendix A Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Subjects must be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria:

* 1. Pregnant or nursing women or subjects expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg [> 10 mg] daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment. Use of inhaled or topical steroids or systemic corticosteroids < 10 mg is permitted.

  2. Prior monoclonal antibody within 4 weeks before study Day 1 or not recovered (≤ Grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier. Exception to this rule would be use of denosumab.

  3. Participation in any other study in which receipt of an investigational study drug occurred within 28 days or 5 half-lives (whichever is longer) prior to first dose. For investigational agents with long half-lives (eg, 5 days), enrollment prior to the fifth half-life requires medical monitor approval.

  4. Subjects who have received prior immune checkpoint inhibitors (eg, anti-CTLA-4, anti-PD-1, anti-PD-L1, and any other antibody or drug specifically targeting T-cell costimulation) or an IDO inhibitor. Subjects who have received experimental vaccines or other immune therapies should be discussed with the medical monitor to confirm eligibility.

  5. Subjects who have received any anticancer medication or therapy in the 21 days prior to receiving their first dose of study medication or have any unresolved toxicity greater than Grade 1 from previous anticancer therapy, except for stable chronic toxicities that are not expected to resolve (ie, peripheral neurotoxicity, alopecia, fatigue, etc).
* Subjects who have had prior radiotherapy within 2 weeks of therapy. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week wash out is permitted for palliative radiation to non-CNS disease with medical monitor approval.Subjects who have any active or inactive autoimmune disease or syndrome (ie, rheumatoid arthritis, lupus, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

Note: Exceptions include subjects with vitiligo or resolved childhood asthma/atopy, hypothyroidism stable on hormone replacement, controlled asthma, Type I diabetes, Graves' disease, or Hashimoto's disease, or with medical monitor approval.

* If subject received major surgery, then they must have recovered adequately from toxicities and/or complications from the intervention prior to starting therapy.
* Patients must have received anticoagulating agent for at least 6 months for any new DVT/PE or other evidence of venous thromboembolism. Patients with evidence of arterial clot must be stable for 3 months on anti-platelet therapy or other anticoagulation as deemed necessary by the investigator.
* Known second primary malignancy that is progressing or requires active treatment. Exceptions include early stage cancers treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 8 weeks before the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases confirmed by repeat imaging, and have not required steroids for at least 14 days before study treatment.
* Evidence of interstitial lung disease or active, history of noninfectious pneumonitis including symptomatic, and/or pneumonitis requiring treatment. Active infection requiring systemic therapy.
* Presence of a gastrointestinal condition that may affect drug absorption.
* Known history of human immunodeficiency virus (HIV; HIV 1/2 antibodies).
* Subject has a known history of or is positive for hepatitis B (HBsAg reactive) or hepatitis C antibody is detected).
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Subjects receiving MAOIs or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening. See Appendix B for prohibited medications associated with MAO inhibition.
* Any history of Serotonin Syndrome (SS) after receiving serotonergic drugs.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful for an unstable cardiovascular event. Screening QTcF interval > 480 milliseconds is excluded. In the event that a single QTcF is > 480 milliseconds, the subject may enroll if the average QTcF for the 3 ECGs is < 480 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the JTc interval may be used in place of the QTcF with sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of the QTcF. Subjects with left bundle branch block are excluded.

Note: QTcF prolongation due to pacemaker may enroll if the JTc is normal.

* Use of any UGT1A9 inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
* History of organ transplant that requires use of immunosuppressive therapy.
* Any condition, including psychiatric conditions, which would jeopardize the safety of the subject or compliance with the Protocol.
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy.
* Known allergy or reaction to any component of either study drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Response (RR) rate | 6 months
  RR defined as patients with complete or partial response as assessed by RECIST v1.1
6 month progression free survival | 6 months
  Percentage of patients without progression of disease or termination of treatment within 6 months of day 1 cycle 1
Response rate with microsatellite instability | 6 months
  RR defined as patients with complete or partial response as assessed by RECIST v1.1
6 months survival in patients with microsatellite instability | 6 months
  Percentage of patients without progression of disease or termination of treatment within 6 months of cycle 1 day 1

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events due to combination of drugs | 2 years
  Percentage of patients with adverse events measured by changes in echocardiogram
Incidence of treatment-emergent adverse events due to combination of drugs | 2 years
  Percentage of patients with adverse events measured by clinical laboratory blood tests
Incidence of treatment-emergent adverse events due to combination of drugs | 2 years
  Percentage of patients with adverse events measured by clinical laboratory urine tests

OTHER OUTCOMES:
Overall survival | 3 years
  Time from the date of starting treatment to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States